CLINICAL TRIAL: NCT03306069
Title: Low-volume Aerobic Interval Training in Overweight Individuals at Increased Cardiometabolic Risk: Impact of Training Intensity on Cardiorespiratory Fitness, Cardiometabolic Risk Profile and Exercise Adherence
Brief Title: Effects of Low-volume Aerobic Interval Training in Overweight Individuals at Increased Cardiometabolic Risk
Acronym: BELITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BELITA-Study
Record Dates: First submitted 2017-09-27; First posted 2017-10-10 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Overweight and Obesity; Metabolic Syndrome
Keywords: Aerobic exercise; Interval training; VO2max; Health Promotion; Inflammation; Body Composition
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Inflammation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment parallel-group, randomized-controlled study
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors involved in data analysis will not be aware of the arm to which the participants were allocated (single-blinded masking).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Experimental): Nutritional therapy / no exercise
  Interventions: Other: Control
- HIIT (Experimental): High-intensity interval training (HIIT) at 90% heart rate maximum (HRmax) combined with Nutritional therapy
  Interventions: Other: HIIT
- MIIT-HR (Experimental): Heart rate based moderate-intensity interval training (MIIT-HR) at 70% heart rate maximum (HRmax) combined with Nutritional therapy
  Interventions: Other: MIIT-HR
- MIIT-LT (Experimental): Lactate threshold based moderate-intensity interval training (MIIT-LT) at 105% of lactate threshold (corresponding ~70-75% HRmax) combined with Nutritional therapy
  Interventions: Other: MIIT-LT

INTERVENTIONS:
Other: Control — Individualized, weight-reducing nutritional therapy and counseling, during a study period of 12 weeks
  Arms: Control
Other: HIIT — Procedures: Nutritional therapy (individualized, weightreducing nutritional therapy and counseling) during a study period of 12 weeks combined with supervised ergometer-based high-intensity interval training (HIIT).
  HIIT:
  * 2 sessions per week
  * 5x1 min at 80-95% HRmax
  * time-effort per week: ~30 min
  Arms: HIIT
Other: MIIT-HR — Procedures: Nutritional therapy (individualized, weightreducing nutritional therapy and counseling) during a study period of 12 weeks combined with supervised ergometer-based moderate-intensity interval training on the basis of HRmax (MIIT-HR).
  MIIT-HR:
  * 2 sessions per week
  * 5x1 min at 65-79% HRmax
  * time-effort per week: ~30 min
  Arms: MIIT-HR
Other: MIIT-LT — Procedures: Nutritional therapy (individualized, weightreducing nutritional therapy and counseling) during a study period of 12 weeks combined with supervised ergometer-based moderate-intensity interval training on the basis of lactate threshold (MIIT-LT).
  MIIT-LT:
  * 2 sessions per week
  * session 1: 2x4 min / session 2: 5x1 min, each at 105% LT
  * time-effort per week: ~30 min
  Arms: MIIT-LT

SUMMARY:
The main purpose of this study is to compare the impact of aerobic interval training intensity on exercise adherence and changes in cardiorespiratory fitness, cardiometabolic risk profile, body composition, inflammatory markers and subjective health outcomes after a 12-week intervention trial in overweight individuals at increased cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >/=30
* presence of at least 2 cardiometabolic risk factors

Exclusion Criteria:

* Healthy persons or patients under age
* Overweight persons without any additional cardiometabolic risk factors
* Pregnancy, Lactation
* Psychological disorders, epilepsy, sever neurological disorders
* Participation in other exercise- or nutrition studies within the last 6 months
* acute cardiovascular disease
* malignant disease
* Electronic implants (defibrillator, pacemaker)
* Persons in mental hospitals by order of authorities or jurisdiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness (CRF) | 12 weeks (baseline to 12 week follow-up assessment)
  CRF will be assessed by measuring Maximum Oxygen uptake (VO2max)

SECONDARY OUTCOMES:
Metabolic Syndrome Z-Score (MetS-Z-Score) | 12 weeks (baseline to 12 week follow-up assessment)
  MetS-Z-Score will be calculated from each individual's measures of waist circumference, mean arterial blood pressure, triglycerides, and HDL-cholesterol, based on equations specific to sex.
Body Composition | 12 weeks (baseline to 12 week follow-up assessment)
  Muscle mass, fat mass and body water will be measured by Bioelectrical Impedance Analysis (BIA)
Insulin sensitivity | 12 weeks (baseline to 12 week follow-up assessment)
  Insulin sensitivity will be estimated using homeostasis model assessment index (HOMA)
Inflammation | 12 weeks (baseline to 12 week follow-up assessment)
  Inflammation will be assessed by measuring levels of inflammatory blood markers
Health-related quality of life | 12 weeks (baseline to 12 week follow-up assessment)
  Health-related quality of life will be assessed by using the standardized and validated EQ-5D-5L Questionnaire
Pain scores | 12 weeks (baseline to 12 week follow-up assessment)
  Pain scores will be assessed by using the standardized and validated Chronic Pain Grade Questionnaire (CPGQ)
Perceived stress | 12 weeks (baseline to 12 week follow-up assessment)
  Perceived stress will be assessed by using the standardized and validated Perceived Stress Questionnaire (PSQ)
Subjective work ability | 12 weeks (baseline to 12 week follow-up assessment)
  Subjective work ability will be assessed by using the standardized and validated Work Ability Index Questionnaire (WAI)

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Reljic, Dr., Principal Investigator — University Erlangen Nuremberg Medical School; Yurdaguel Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports,, Erlangen, Germany

REFERENCES:
- [Derived] Reljic D, Frenk F, Herrmann HJ, Neurath MF, Zopf Y. Low-volume high-intensity interval training improves cardiometabolic health, work ability and well-being in severely obese individuals: a randomized-controlled trial sub-study. J Transl Med. 2020 Nov 7;18(1):419. doi: 10.1186/s12967-020-02592-6. PMID 33160382